CLINICAL TRIAL: NCT02120898
Title: A Multicenter, Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Comparison Study to Determine the Therapeutic Equivalence of Generic Imiquimod Cream, 2.5% and Zyclara® (Imiquimod) Cream, 2.5% in Subjects With Actinic Keratoses
Brief Title: A Study to Evaluate the Safety and Efficacy Imiquimod Cream, 2.5% in Participants With Actinic Keratoses
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 094-3153-301
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; Imiquimod; Zyclara
MeSH Terms: conditions — Keratosis, Actinic | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Generic Imiquimod Cream 2.5% (Experimental): Generic imiquimod cream 2.5% will be applied once daily approximately 1 to 2 hours before bedtime to the skin of the treatment area (either full face [excluding the ears] or balding scalp) for two, 2-week treatment cycles separated by a 2-week no-treatment period. Participants will apply test article for 14 consecutive days for each treatment cycle.
  Interventions: Drug: Imiquimod
- Zyclara® (Imiquimod) Cream 2.5% (Active Comparator): Zyclara® (imiquimod) cream 2.5% will be applied once daily approximately 1 to 2 hours before bedtime to the skin of the treatment area (either full face [excluding the ears] or balding scalp) for two, 2-week treatment cycles separated by a 2-week no-treatment period. Participants will apply test article for 14 consecutive days for each treatment cycle.
  Interventions: Drug: Zyclara®
- Vehicle Cream (Placebo Comparator): Vehicle cream will be applied once daily approximately 1 to 2 hours before bedtime to the skin of the treatment area (either full face [excluding the ears] or balding scalp) for two, 2-week treatment cycles separated by a 2-week no-treatment period. Participants will apply test article for 14 consecutive days for each treatment cycle.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: Imiquimod — Cream, generic formulation of the brand product.
  Arms: Generic Imiquimod Cream 2.5%
Drug: Zyclara® — Cream, brand product.
  Arms: Zyclara® (Imiquimod) Cream 2.5%
Drug: Vehicle Cream — Vehicle cream in the same image of the generic imiquimod. Has no active ingredient.
  Arms: Vehicle Cream

SUMMARY:
The purpose of this study it so compare the safety and efficacy profiles of a generic imiquimod 2.5% cream to the reference listed Zyclara® (imiquimod) cream in the treatment of actinic keratosis (AK).

DETAILED DESCRIPTION:
Aldara® (imiquimod) Cream, 5% was the first imiquimod product approved by the Food and Drug Administration (FDA) for the topical treatment of AK, superficial basal cell carcinoma and external genital and perianal warts. The FDA approved regimen for the treatment of AK is application of 250 milligrams (mg) of cream twice a week for 16 weeks to a 25 square centimeters (cm^2) area. In 2011, a lower strength imiquimod cream, Zyclara (imiquimod) Cream, 2.5% was approved by the FDA. When used for the treatment of AK, Zyclara is applied for a shorter duration and in an expanded treatment area (for example, face or scalp) in comparison to Aldara®. This study will be conducted in compliance with the protocol, Good Clinical Practice (GCP) and the applicable regulatory requirement(s). Marketed by Medicis, Zyclara® (imiquimod) cream 2.5% is a safe and effective topical therapy for the treatment of AK of the face and scalp. Actavis has developed a generic formulation of imiquimod 2.5% cream and the current study is designed to evaluate the safety and efficacy of this formulation.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a male or female, 18 years of age or older.
* Participant has provided written informed consent.
* Participant is willing and able to apply the test article as directed, comply with study instructions and commit to all follow-up visits for the duration of the study.
* Participant has a clinical diagnosis of AK with at least 5 and no more than 20 clinically typical, visible or palpable AK lesions, each at least 4 millimeters (mm) in diameter, in an area greater than 25 cm^2 on the face (excluding ears) or balding scalp, but not both.
* Participant is in good general health and free of any disease state or physical condition that might impair evaluation of AK lesions or which, in the investigator's opinion, exposes the participant to an unacceptable risk by study participation.
* Females must be post-menopausal, surgically sterile or use an effective method of birth control, with a negative urine pregnancy test (UPT) at the Baseline visit.

Exclusion Criteria:

* Participant is pregnant, lactating, or is planning to become pregnant during the study.
* Participant has hyperkeratotic, hypertrophic or atypical AKs (for example, AK greater than [>] 1 cm^2 in size) in the treatment area.
* Participant is currently enrolled in an investigational drug or device study.
* Participant plans to be exposed to artificial tanning devices or excessive sunlight during the trial.
* Participant is immunosuppressed (for example; human immunodeficiency virus [HIV], systemic malignancy, graft vs. host disease, etc.).
* Participant has experienced an unsuccessful outcome from previous imiquimod therapy (an unsuccessful outcome is defined as after a reasonable therapeutic trial with no compliance issues and the topical drug do not work).
* Participant has used an investigational drug or investigational device within 30 days prior to the Baseline visit.
* Participant has had dermatologic procedures or surgeries such as: laser resurfacing, PUVA (Psoralen + ultraviolet A) therapy, UVB therapy, chemical peels or dermabrasion on the face or balding scalp within 6 months prior to the Baseline visit.
* Participant has cryodestruction or chemodestruction, curettage, photodynamic therapy, surgical excision or other treatments for AK on the designated treatment area (face or scalp) within 1 month prior to the Baseline visit.
* Participant has used oral corticosteroid therapy, interferon, cytotoxic drugs, immunomodulators, immunosuppressive therapies or retinoids within 1 month prior to the Baseline visit.
* Participant has used topical medications; corticosteroids, alpha hydroxyl acids (for example; glycolic acid, lactic acid etc. >5%), beta hydroxy acid (salicylic acid >2%), urea >5%, 5-fluorouracil, diclofenac, imiquimod, ingenol mebutate or prescription retinoids (for example; tazarotene, adapalene, tretinoin) to the face or balding scalp within one month prior to the Baseline visit.
* Participant has used topical creams, lotions or gels of any kind to the selected treatment area within one day prior to the Baseline visit.
* Participant has lesions suspicious for skin cancer (skin cancer not ruled out by biopsy) or untreated skin cancers within the selected treatment area (face or scalp).
* Participant has a history of sensitivity to any of the ingredients in the test articles.
* Participant has any skin pathology or condition (for example; facial/scalp psoriasis, atopic dermatitis, acne, rosacea, etc.) that, in the investigator's opinion, could interfere with the evaluation of the test article, worsen due to the treatment or requires the use of interfering topical, systemic or surgical therapy.
* Participant has any condition which, in the investigator's opinion, would make it unsafe or precludes the participant's ability to fully participate in this research study.
* Participant is known to be noncompliant or is unlikely to comply with the requirements of the study protocol (for example; due to alcoholism, drug dependency, mental incapacity) in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2013-10-10 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2014-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Actavis Inc.
Locations (27):
- United States (27):
  - Site 1, Birmingham, Alabama
  - Site 10, Fremont, California
  - Site 8, Los Angeles, California
  - Site 24, Denver, Colorado
  - Site 28, Boca Raton, Florida
  - Site 26, Brandon, Florida
  - Site 27, Brandon, Florida
  - Site 21, Boise, Idaho
  - Site 3, Arlington Heights, Illinois
  - Site 17, Champaign, Illinois
  - Site 7, Carmel, Indiana
  - Site 15, Indianapolis, Indiana
  - Site 22, Plainfield, Indiana
  - Site 23, South Bend, Indiana
  - Site 16, Clinton Township, Michigan
  - Site 13, Fridley, Minnesota
  - Site 9, Albuquerque, New Mexico
  - Site 4, High Point, North Carolina
  - Site 11, Wilmington, North Carolina
  - Site 18, Winston-Salem, North Carolina
  - Site 25, Portland, Oregon
  - Site 20, Fountain Inn, South Carolina
  - Site 6, Knoxville, Tennessee
  - Site 5, Nashville, Tennessee
  - Site 14, Austin, Texas
  - Site 12, College Station, Texas
  - Site 2, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 467 participants were enrolled and randomized in 2:2:1 to receive generic imiquimod cream 2.5%, zyclara® (imiquimod) cream 2.5%, or vehicle cream.
Groups:
- Generic Imiquimod Cream 2.5%: Generic imiquimod cream 2.5% was applied once daily approximately 1 to 2 hours before bedtime to the skin of the treatment area (either full face [excluding the ears] or balding scalp) for two, 2-week treatment cycles separated by a 2-week no-treatment period. Participants applied test article for 14 consecutive days for each treatment cycle.
- Zyclara® (Imiquimod) Cream 2.5%: Zyclara® (imiquimod) cream 2.5% was applied once daily approximately 1 to 2 hours before bedtime to the skin of the treatment area (either full face [excluding the ears] or balding scalp) for two, 2-week treatment cycles separated by a 2-week no-treatment period. Participants applied test article for 14 consecutive days for each treatment cycle.
- Vehicle Cream: Vehicle cream was applied once daily approximately 1 to 2 hours before bedtime to the skin of the treatment area (either full face [excluding the ears] or balding scalp) for two, 2-week treatment cycles separated by a 2-week no-treatment period. Participants applied test article for 14 consecutive days for each treatment cycle.
Period: Overall Study
Arm/Group | Generic Imiquimod Cream 2.5% | Zyclara® (Imiquimod) Cream 2.5% | Vehicle Cream
Started | 187 | 187 | 93
Safety Population (All randomized participants who received study drug.) | 187 | 187 | 93
Intent-to-Treat (ITT) Population (Applied at least 1 dose of study drug, and returned for at least 1 post-baseline evaluation.) | 183 | 185 | 93
Completed | 178 | 181 | 89
Not Completed | 9 | 6 | 4
Not completed — Withdrawal by Subject | 4 | 2 | 2
Not completed — Non-compliance with study drug | 3 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 1
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Generic Imiquimod Cream 2.5% | Zyclara® (Imiquimod) Cream 2.5% | Vehicle Cream | Total
Number analyzed (Participants) | 187 | 187 | 93 | 467
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (9.15) | 66.1 (9.82) | 67.2 (9.85) | 66.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 14 | 56
  Male | 168 | 164 | 79 | 411

OUTCOME MEASURES:

1. Primary Outcome: Complete Clearance Rate - Percentage of Participants With Treatment Success: Per-Protocol (PP) Population
Description: Complete clearance rate (treatment success) was defined as the percentage of participants in each treatment group with a count of zero actinic keratosis (AK) lesions in the treatment area at Week 14. All AKs (baseline and new lesions) independent of size within the treatment area were included in the efficacy lesion count. The AK clearance rate for a participant was calculated as follows: {1 - [ (number of AK lesions at Week 14) / (number of AK lesions at Baseline)]} * 100.
Time Frame: Week 14
Population: PP population, a subset of intent-to-treat (ITT) population (all randomized participants who applied at least 1 dose of study drug, and returned for at least 1 post-baseline evaluation) included participants who met all entry criteria, complaint with study drug and completed Week 14 evaluation with no protocol violation.
Measure: Number; unit: percentage of participants
Arm/Group | Generic Imiquimod Cream 2.5% | Zyclara® (Imiquimod) Cream 2.5% | Vehicle Cream
Number analyzed (Participants) | 161 | 162 | 83
percentage of participants | 12.4 | 13.6 | 4.8
Statistical Analysis 1: Comparison: Generic Imiquimod Cream 2.5% vs Zyclara® (Imiquimod) Cream 2.5%; Analysis was performed using 90% Wald's confidence interval (CI) with a continuity correction or the difference (generic imiquimod - Zyclara) in complete clearance rates; Test type: Equivalence — 90% CI interval was -0.20 to +0.20 for therapeutic equivalence; p = 0.0702, Fisher Exact; Percentage difference = -1.16, 90% CI 2-sided [-7.93 to 5.62]

2. Primary Outcome: Complete Clearance Rate - Percentage of Participants With Treatment Success: ITT Population
Description: Complete clearance rate (treatment success) was defined as the percentage of participants in each treatment group with a count of zero AK lesions in the treatment area at Week 14. All AKs (baseline and new lesions) independent of size within the treatment area were included in the efficacy lesion count. The AK clearance rate for a participant was calculated as follows: {1 - [ (number of AK lesions at Week 14) / (number of AK lesions at Baseline)]} * 100.
Time Frame: Week 14
Population: ITT population included all randomized participants who applied at least 1 dose of study drug, and returned for at least 1 post-baseline evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Generic Imiquimod Cream 2.5% | Zyclara® (Imiquimod) Cream 2.5% | Vehicle Cream
Number analyzed (Participants) | 183 | 185 | 93
percentage of participants | 12.6 | 12.4 | 4.3
Statistical Analysis 1: Comparison: Generic Imiquimod Cream 2.5% vs Zyclara® (Imiquimod) Cream 2.5%; Analysis was performed using 90% Wald's CI with a continuity correction or the difference (generic imiquimod - Zyclara) in complete clearance rates; Test type: Superiority; p = 0.0318, Fisher Exact — Threshold for significance at 0.05 level; Percentage difference = 0.14, 90% CI 2-sided [-6.08 to 6.35]

3. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Mild AEs: awareness of sign or symptom, but easily tolerated. Moderate AEs: discomfort sufficient to cause interference with normal activities. Severe AEs: inability to carry out usual activities. Serious AEs: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline (Day 1) up to Week 14
Population: Safety population included all randomized participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Generic Imiquimod Cream 2.5% | Zyclara® (Imiquimod) Cream 2.5% | Vehicle Cream
Number analyzed (Participants) | 187 | 187 | 93
Participants
  Any AEs | 51 | 50 | 22
  Any AEs in treatment area | 7 | 5 | 5
  SAEs | 6 | 4 | 2
  SAEs in treatment area | 0 | 0 | 1
  Mild AEs | 31 | 29 | 10
  Moderate AEs | 16 | 20 | 11
  Severe AEs | 4 | 1 | 1

4. Secondary Outcome: Number of Participants With Local Skin Reactions
Description: Local skin reactions included erythema, flaking/scaling/dryness, scabbing/crusting, pruritus, erosion/ulceration, pain, edema, and weeping/exudate. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline (Day 1) up to Week 14
Population: Safety population included all randomized participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Generic Imiquimod Cream 2.5% | Zyclara® (Imiquimod) Cream 2.5% | Vehicle Cream
Number analyzed (Participants) | 187 | 187 | 93
Participants
  Erythema | 33 | 30 | 17
  Flaking/Scaling/Dryness | 32 | 29 | 22
  Scabbing/Crusting | 22 | 13 | 11
  Pruritus | 12 | 5 | 4
  Erosion/Ulceration | 3 | 2 | 1
  Pain | 2 | 2 | 0
  Edema | 2 | 2 | 0
  Weeping/Exudate | 1 | 1 | 0

5. Other Pre Specified Outcome: Percentage of Drug Compliance
Description: The overall drug compliance (%) = (Observed Consumption / Expected Consumption) * 100%.
Time Frame: Baseline (Day 1) up to Week 6
Population: ITT population included all randomized participants who applied at least 1 dose of study drug, and returned for at least 1 post-baseline evaluation. Here 'Overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of drug compliance
Arm/Group | Generic Imiquimod Cream 2.5% | Zyclara® (Imiquimod) Cream 2.5% | Vehicle Cream
Number analyzed (Participants) | 182 | 183 | 93
percentage of drug compliance | 96.55 (10.233) | 97.83 (7.653) | 97.43 (9.410)

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to Week 14
Description: Safety population included all randomized participants who received study drug.
Arm/Group | Generic Imiquimod Cream 2.5% | Zyclara® (Imiquimod) Cream 2.5% | Vehicle Cream
Serious Adverse Events (participants affected / at risk) | 6/187 | 4/187 | 2/93
Other Adverse Events (participants affected / at risk) | 16/187 | 15/187 | 7/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Generic Imiquimod Cream 2.5% (N=187) | Zyclara® (Imiquimod) Cream 2.5% (N=187) | Vehicle Cream (N=93)
Autoimmune disorder (Immune system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Generic Imiquimod Cream 2.5% (N=187) | Zyclara® (Imiquimod) Cream 2.5% (N=187) | Vehicle Cream (N=93)
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 0
Application site pain (General disorders) | 4 | 1 | 0
Fatigue (General disorders) | 1 | 4 | 0
Nasopharyngitis (Infections and infestations) | 5 | 0 | 2
Sinusitis (Infections and infestations) | 3 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 5 | 5 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.

DOCUMENTS (2):
  • Study Protocol (2013-07-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT02120898/Prot_000.pdf
  • Statistical Analysis Plan (2014-04-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT02120898/SAP_001.pdf